CLINICAL TRIAL: NCT06044220
Title: Evaluation of the Effectiveness of Testicular Self-examination Training Given to Male University Students
Brief Title: Testicular Self-examination Training Given to Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Öznur KIRMIZI AY, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OKIRMIZIAY-001
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Testicular Neoplasm
Keywords: Testicular Cancer; Testicular self-exam; Planned behavior theory scale
MeSH Terms: conditions — Testicular Neoplasms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group is given a 3-month reminder after the TSE training.
  Interventions: Behavioral: Intervention
- control (Other): No training or reminders are given to the control group
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention — The intervention group was given training on male reproductive health and testicular self-examination after the pretest. Posttest was administered after the training. He was reminded to perform TSE for 3 months after the training. After the reminders, a follow-up test was applied.
  Arms: Intervention
Other: Control — Pretest and posttest were administered to the control group at the same time as the intervention group. After reminding the intervention group to perform TSI for 3 months, a follow-up test was performed in the control group.
  Arms: control

SUMMARY:
The aim of this quasi-experimental control group study was to evaluate the effectiveness of testicular self-examination training given to male university students.

Hypotheses; H1a: Immediately after the training and three months after the training, the experimental and control groups' Planned Behavior Theory scale intention sub-dimension scores related to Testicular Self-Examination will increase.

H1b: Immediately after the training and three months after the training, the experimental and control groups' Planned Behavior Theory scale attitude sub-dimension scores related to Testicular Self-Examination will increase.

H1c: Immediately after the training and three months after the training, the experimental and control groups' Planned Behavior Theory scale subjective norm sub-dimension scores on Testicular Self-Examination will increase.

H1d: Immediately after the training and three months after the training, the experimental and control groups' Planned Behavior Theory scale perceived behavioral control sub-dimension scores will increase.

H1e: Immediately after the training and three months after the training, the scores of the Planned Behavior Theory scale self-efficacy sub-dimension related to Testicular Self-Examination will increase in the experimental and control groups.

H1f: Immediately after the training and three months after the training, the experimental and control group's Planned Behavior Theory scale total scores on Testicular Self-Examination will increase.

A questionnaire will be administered to the participants before and after the training of male health promotion and testicular self-examination, and the retest will be filled after the reminders about the smallpox given for 3 months.

The researcher will compare the intervention and control group to see if the behavior of performing testicular self-examination regularly occurs.

DETAILED DESCRIPTION:
The data of the research were obtained from the students of Medical Documentation and Secretarial Program, Medical Promotion and Marketing Program and Optician Program affiliated to Bartın University Vocational School of Health Services Medical Services and Techniques Department between 27 December - 5 April 2022. The research was carried out in 3 stages.

pre-enterprise phase; Data collection forms were applied to n=102 participants who met the inclusion criteria and accepted the study (pretest). One participant with varicocele and one participant with a history of undescended testicles were excluded from the study. Experiment (n=51) and control (n=49) groups were formed by drawing lots between the primary and secondary education programs.

Initiative stage; The "Male Health Promotion Training Program for Self-Testicular Examination" prepared by the researcher as a result of literature review (Power, et al. 2021; Taylor, 2004), was carried out in two sessions on different days in the same week. In the first session (30 minutes), the Anatomy of Male Reproductive Organs, Testicular Cancer and Risky Situations Caused by Testicular Cancer, in the second session (30 minutes) Testicular Self-Examination, the Importance of Regular Testicular Examination, and Fields of Expertise in Suspicion of Testicular Cancer were discussed. Data collection forms were applied for the second time immediately after the intervention (posttest). After the intervention, once a month for 3 months, the participants in the experimental group were reminded via mobile phone with the question "Have you done your Testicular Self Examination this month?".

Post-intervention stage; At the end of the third month after the intervention, the data collection forms were applied again and the research process was completed (Follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Being a continuous student at Vocational School of Health Services,
2. Being over 18 years of age,
3. Volunteering.

Exclusion Criteria:

1. Those with a history of TC,
2. Those with a family history of TC and
3. Those with a history of testicular surgery such as undescended testicles, varicocelectomy and hydrocelectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
survey form and Theory of Planned Behavior scale for testicular self-examination | one week
  A survey form consisting of 21 questions, prepared by the researcher by reviewing the literature, and the Theory of Planned Behavior scale adapted to Turkish on Testicular Self-Examination were applied as a pretest.

SECONDARY OUTCOMES:
Planned behavior theory scale related to testicular self-examination | one week
  The Theory of Planned Behavior Scale on Testicular Self-Examination was applied as a posttest.
  The minimum score to be obtained from the scale is 16 and the maximum is 112. Each dimension of the scale is evaluated separately, and as the score increases, positive behavior increases.

OTHER OUTCOMES:
Theory of Planned Behavior scale for testicular self-examination | three months
  The Theory of Planned Behavior Scale on Testicular Self-Examination was applied as a follow-up test.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan KAR ŞEN, Study Director — Assist. Prof. Dr., Department of Nursing Sciences
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No